CLINICAL TRIAL: NCT04307342
Title: Posterior MIPO for Humerus Diaphyseal Fractures With Extra-articular Distal Humeral Anatomical Plate
Brief Title: Posterior Minimally Invasive Plate Osteosynthesis (MIPO) for Humerus Diaphyseal Fractures
Acronym: MIPOH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Traumatologico Dr. Teodoro Gebauer Weisser (Other)
Collaborators: University of Chile (Other)
Responsible Party: Principal Investigator, Julio Contreras, Shoulder and Elbow Surgeon, Instituto Traumatologico Dr. Teodoro Gebauer Weisser
Other Study IDs: MIPOH
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Humerus Fracture
Keywords: humerus; fracture; osteosynthesis
MeSH Terms: conditions — Humeral Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Posterior MIPO: Patients treated with posterior MIPO for Humerus Diaphyseal Fractures With Extra-articular Distal Humeral Anatomical Plate
  Interventions: Procedure: MIPO with Extra-articular Distal Humeral Anatomical Plate

INTERVENTIONS:
Procedure: MIPO with Extra-articular Distal Humeral Anatomical Plate — MIPO with Extra-articular Distal Humeral Anatomical Plate

SUMMARY:
The primary objective is to evaluate the clinical, functional and radiological results in patients treated with posterior MIPO for Humerus Diaphyseal Fractures With Extra-articular Distal Humeral Anatomical Plate.

DETAILED DESCRIPTION:
The primary objective is to evaluate the clinical, functional and radiological results in patients treated with posterior MIPO for Humerus Diaphyseal Fractures With Extra-articular Distal Humeral Anatomical Plate.

Clinical

* Pain
* ROM

Functional

* Constant Score
* MEPS
* QuickDASH

Radiological

- Bone union

Complications

* Infection
* Nerve injury

ELIGIBILITY:
Inclusion Criteria:

* Closed diaphyseal humerus fracture at the junction of the middle third with distal

Exclusion Criteria:

* Open fractures, proximal humerus extension, distal articular compromise, polytrauma, more than 2 weeks of trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in the emergency department of the Instituto Traumatológico for a fracture of the humerus
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Bone union | 6 months
  Radiological Bone union (X-ray or CT)

SECONDARY OUTCOMES:
Pain (Quantity) | 1 month, 6 months, 1 year
  Visual Analog Scale
Range of Motion (Degrees of flexion, extension, pronation and supination) | 1 month, 6 months, 1 year
  Physical Exam
Constant Score | 1 month, 6 months, 1 year
  Score
Mayo Elbow Score | 1 month, 6 months, 1 year
  Score
Quick Disabilities of the Arm, Shoulder and Hand | 1 month, 6 months, 1 year
  Score
Radial nerve injury | 1 month, 6 months, 1 year
  Physical exam (electromyography when needed)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Traumatológico, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF, CSR